CLINICAL TRIAL: NCT04122482
Title: A Randomized Controlled Trial of an Online Psychoeducation Course for Improving Knowledge and Access to Mental Health Accommodations in Canadian Enterprises
Brief Title: An Online Course for Improving Knowledge and Access to Mental Health Accommodations in Canadian Enterprises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2019-126
Record Dates: First submitted 2019-09-23; First posted 2019-10-10 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2021-10

CONDITIONS: Depression, Anxiety
Keywords: Mental health accommodation; Canadian buisness; Psychoeducation; ICBT
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Factorial Assignment Factor 1: Receive course material immediately Factor 2: Receive course material in 8 weeks
  Each client will be randomized to one of two conditions:
  Condition 1: They receive access to the course material immediately. Condition 2: They receive access to the course material after 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): In this arm, participants will be given access to the course material shortly after eligibility criteria is confirmed. They will be asked to complete post-measures questionnaires at 4 weeks and 8 weeks following completion of the course material.
  Interventions: Behavioral: Psychoeducation Course
- Wait-list Control (Experimental): In this arm, participants will be given access to the course material 8 weeks following confirmation of their eligibility. During, the 8-week waiting period they will be asked to complete questionnaires at 4 weeks and 8 weeks. At 8 weeks they will be given access to the course material and will be asked to complete the same questionnaires 4- and 8-weeks following completion of the course material.
  Interventions: Behavioral: Psychoeducation Course

INTERVENTIONS:
Behavioral: Psychoeducation Course — The investigators are assessing the efficacy of the accommodations course. Specifically, the investigators will evaluate the impact on requesting and receiving accommodations for anxiety and/or depression, employee knowledge of accommodations, and employee self-stigmatizing attitudes. The investigators will also assess if the course helps improve comfort level of disclosing a mental health diagnosis and rates of disclosure in the workplace.
  Other Names: Wait-list Control

SUMMARY:
Available research on mental health accommodations within the workplace suggests that employees with mental health concerns require accommodations (e.g., flexible scheduling, quiet spaces), but only a fraction of employees will receive the accommodations they have requested. Reported barriers to receiving mental health accommodations include concerns regarding stigma, lack of knowledge about appropriate accommodations, financial constraints of the employer, and size of the organization. While there is growing research on workplace accommodations, there is a paucity of research available on interventions aimed at improving accommodation usage, particularly within SMEs. To address this gap, the intent of the proposed study is to develop and implement an online psychoeducation course to increase employees' accommodation knowledge and usage within Canadian enterprises. Once the course is developed, reviewed, and implemented, an additional aim of the proposed study will be to test the efficacy of the course using a two-arm, randomized controlled trial comparing the intervention to a wait-list control group. A total of 86 participants experiencing workplace impairments due to a depressive and/or anxiety disorder will be randomly assigned to a psychoeducation group or wait-list control group. A 2x3 repeated measures (i.e., pre-course, at four weeks and eight weeks) mixed model ANOVA will be used to analyze the effects of the intervention on accommodation requests, knowledge of accommodations, absenteeism/presenteeism rates, employee self-efficacy, and psychological symptoms. The results of the study may be used to develop future offerings of the course and improve mental health accommodations practices within Canadian enterprises.

DETAILED DESCRIPTION:
In this study, the first phase of the study will be to develop the online psychoeducation course. Once the course is developed it will be reviewed by experts in the field of accommodations (e.g., Human Resource professionals, lawyers) and their suggestions will be reviewed and possibly implemented before the course is delivered to employees. Experts providing feedback will be asked to review and complete a consent form prior to reviewing one or more lessons. After reviewing a lesson, they will be provided with an opportunity to give lesson feedback through the completion of a short questionnaire. Total participation time is expected to be 1 hour. Experts will be eligible for the study if they meet the following criteria: (1) are 18 years of age or older; (2) have knowledge or experience with workplace accommodations; and (3) are Canadian residents. Experts will be excluded if he/she: (1) is not 18 years of age or older); (2) Do not have knowledge or experience with workplace accommodations; (3) are not a resident of Canada

The course will be comprised of the following lessons:

Lesson 1: Anxiety and depression in the workplace. This lesson will include information on how to identify symptoms of depression and anxiety in the workplace. To accomplish this the DSM-5 criteria for depression and anxiety will be provided along with practical work examples (e.g., difficulty with concentration in meetings). Participants will also be presented with examples of the functional limitations that are commonly associated with depression and anxiety symptoms (e.g., missing important deadlines due to procrastination behaviours). Information on the prevalence of depression and anxiety in Canada/World will also be provided to counteract any stigmatic attitudes or beliefs.

Lesson 2: Accommodations for mental health concerns. Within this lesson, participants will be presented with the Canadian legislation on reasonable workplace accommodations. This information will include a discussion on undue hardship and how this may impact the receipt and types of accommodations available within Canadian enterprises. Participants will also be provided with common examples of accommodations frequently identified within the research literature (e.g., flexible work schedules, quiet spaces). In addition, the benefits of receiving accommodations for mental health concerns (e.g., improved productivity, reduced symptomology) will be discussed. The lesson will conclude with the potential barriers (e.g., stigma, organizational barriers) and facilitators (e.g., supportive work environments) to requesting and receiving accommodations. Strategies to overcome potential barriers will also be addressed.

Lesson 3: Requesting an accommodation and disclosure. This lesson will focus on strategies for requesting an accommodation within a Canadian enterprise. This will include information on when, how, to whom, and what should be disclosed when requesting an accommodation. Employees will also be provided with information on the pros and cons of making an accommodation request. In addition, they will be provided with information on what to disclose when making the request (i.e., full disclosure ["I have depression] or selective disclosure ["I have an illness]), the pros and cons of disclosure, and information on the tasks for preparing to disclose. It will also be emphasized within the lesson that full disclosure may not be required to receive an acceptable accommodation.

Lesson 4: Future management. The psychoeducational course will conclude with a lesson on strategies for managing depression and anxiety symptoms within Canadian enterprises with or without an accommodation. This will include information on managing symptoms within the work environment such as, managing expectations, tackling avoidance strategies, progressive muscle relaxation, and fostering workplace relationships/supports.

The second aim of the proposed study will be to test the efficacy of the course using a two arm, randomized controlled trial. The sample size of 43 participants per arm is based on a power analysis for an ANOVA: repeated measures, between factors, with a medium effect size (f = 0.25), an alpha of 0.05, correlation among repeated measure of 0.5, and power of 0.80.

All interested participants will be directed to the study website (www.onlinetherapyuser.ca), where they will be presented with a consent form explaining the screening protocol (i.e., online screening consent). After consent is given, participants will be assessed for program eligibility using an Internet-delivered screening questionnaire. The online screening questionnaire captures demographic information (e.g., sex, ethnicity, location), contact details (e.g., telephone number, email address), eligibility information (e.g., medical history, mental health history, symptom measurements), and information on workplace functioning (e.g., self-reported absenteeism, presenteeism, disclosure questions, self-efficacy, self-stigma, workers' relation scale, workplace inclusion). This data will be made available to participants in an online survey created and hosted by REDcap (Research Electronic Data Capture) software.

Once participants have been assessed for program eligibility using the online screening tool, they will asked to schedule a telephone interview. During the telephone interview, the primary investigator will ask a series of follow-up questions (i.e., Telephone Interview Guide) to the online screening questionnaire to ensure program eligibility as per exclusion criteria. Participants who meet any of the exclusion criteria during the online screening phase will be provided with an explanation for their ineligibility and encouraged to contact the researcher via email if they have any questions or concerns.

Participants who are appropriate for the study will be assigned to their randomized group (i.e., Psycho-education course or wait-list control group). At this point, participants assigned to the psycho-education group will be provided user-names and temporary password words by phone to access the course. Participants assigned to the wait-list group will be provided with their user name and password 8 weeks following the telephone screening date. Before beginning the course, all participants will be presented with a course consent form that will explain the nature of the intervention.

The lessons will take approximately 30 to 45 minutes for participants to review. Once participants have completed a lesson, they will be granted access to the next lesson the following day, which will allow them to complete multiple lessons within any given week. To minimize time pressures, participants will be instructed that follow-up measures (i.e., same measures included in the screening questionnaire minus the AUDIT/DUDIT and clinical history) will be available four weeks and eight weeks after they have been provided access to the course. Should negative effects be observed (e.g. self-reported symptoms increase, absenteeism/presenteeism numbers significantly rise) at any point, participants will be reminded of the resources (e.g., family doctor, mental health websites, mental health agencies) available to them. These resources will be documented and posted on the website for easy reference.

The use of a wait-list control group will provide a comparison group to determine the effects of the psychoeducation course. It will also circumvent any ethical concerns with failing to provide a potentially helpful intervention. Participants assigned to the wait-list group will be assigned a start date eight weeks after the pre-screen interview and sent an automatic reminder email a few days prior to their start date. The wait-list group will also be sent a link through email to complete measures (i.e., PHQ-9, Accommodation/Disclosure questions, WHO HPQ) four-weeks after the telephone screen for comparison purposes and to maintain engagement in the study. No further contact will be provided during the eight-week wait-list period. Following completion of the wait-list period, the participants will be provided their user name and password so they may access the psycho-education course and measures will be requested again at 4-weeks and 8-weeks post course access.

ELIGIBILITY:
Inclusion Criteria:

* are 18 years of age or older;
* are a resident of Canada;
* are experiencing at least clinically significant symptoms of anxiety and/or depression (i.e., symptoms are severe enough to impact work performance);

  - I.e., a GAD-7 score of 10 or greater, or SIAS score of 7 or greater, SPS-6 score of 2 or greater, PHQ-0 score of 10 or greater, be absent from work a minimum of .3 days in the last 28 days, have a presenteeism score of 40 or greater.
* have not been hospitalized within the last year for mental health and/or suicide risk concerns;
* have access to a secure computer and the Internet, and is comfortable using technology.

Exclusion Criteria:

* are younger than 18 years of age;
* are not a resident of Canada;
* are experiencing minimal or no symptoms of anxiety and/or depression;
* have been hospitalized within the last year for mental health and/or suicide risk concerns;
* have unmanaged problems with alcohol, drugs, psychosis, or mania;
* do not have access to a secure computer and the Internet or is not comfortable using technology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2020-11-21 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Assessing change of requesting and/or receiving accommodations between course start date and 8 weeks post course completion. | 8 weeks
  We will be assessing the impact of the psychoeducation course on requesting and/or receiving workplace accommodations for anxiety and/or depression symptoms. This will be assessed using a questionnaire, which will include questions such as "Have you ever requested from your current company any change or accommodation in your job or workplace to better meet your mental health needs?" This questionnaire includes dichotomous questions (yes/no) and there is one scale that asks how comfortable participants are requesting an accommodation (min: 1; max: 10). A higher value represents more comfort requesting an accommodation.
Efficacy of online psychoeducation course on self-stigmatizing attitudes as measured by Self-stigma of Mental Illness Scale - Short Form (SSMIS-SF) | 8 weeks
  We will be assessing the impact of the psychoeducation course on employees' self-stigmatizing attitudes. The investigators will be assessing 4 sub-scales (Aware, Agree, Apply, and Hurts Self). Each sub-scale has the following minimum and maximum values Min: 5 Max: 45 Higher values represent more self-stigmatizing attitudes.
Assessing change in employee knowledge of accommodations between course start date and 8 weeks post course completion | 8 weeks
  We will be assessing employees' knowledge of accommodations before and after receiving the course material. This will be assessed using a questionnaire that includes likert scales and open-ended questions such as "On a scale from 1 to 10, where 1 is "no knowledge" and 10 is "very knowledgeable how much do you know about workplace accommodations for mental health conditions?" and "Please list the accommodations you are comfortable requesting?"
Impact of receiving accommodations on absenteeism and presenteeism rates as measured by the World Health and Work Performance Questionnaire (WHO-HPQ). | 8 weeks
  Change in absenteeism and presenteeism rates in terms of the total number of missed work days or lower productivity days during the previous 28 days.
Impact of receiving accommodations on employee self-efficacy as measured by New General Self-Efficacy Scale (NGSE). | 8 weeks
  Change in employees' self-efficacy scores during the previous 4 weeks. The total score is calculated by total score for each participant and taking the average rating of the items selected.
  Minimum score: 1 Maxium score: 5 Lower values represent lower self-efficacy
Impact of receiving accommodations on employee symptom severity as measured bygeneral anxiety measures (GAD-7) | 8 weeks
  Change in employees' self-reported symptom severity during the previous 4 weeks.
  GAD-7- Min score = 0; Max score = 21 - Higher scores represents more severe symptoms
Impact of receiving accommodations on employee symptom severity as measured by social interaction anxiety measures (SIAS-6). | 8 weeks
  Change in employees' self-reported symptom severity during the previous 4 weeks.
  SIAS-6: Min score = 0; Max score = 24 - Higher scores represents more severe symptoms
Impact of receiving accommodations on employee symptom severity as measured by social phobia anxiety measures (SPS-6). | 8 weeks
  Change in employees' self-reported symptom severity during the previous 4 weeks.
  SPS-6: Min score = 0; Max score = 24 - Higher scores represents more severe symptoms
Impact of receiving accommodations on employee symptom severity as measured by depression measures (PHQ-9) | 8 weeks
  Change in employees' self-reported symptom severity during the previous 4 weeks.
  PHQ-9 - Min score = 0; Max score = 27 - Higher scores represents more severe symptoms
Assessing change in employee relationships within the workplace as measured by the Workplace Relationships Scale (WRS). | 8 weeks
  Change in employees' workplace relationships during the previous 4 weeks.
  WRS scores will range from:
  Min: 9 Max: 63 Higher scores represents more interpersonal conflict at work.
Identification of workplace accommodations received for anxiety and/or depression symptoms. | 8 weeks
  Participants will be asked to list any workplace accommodations they have received for the anxiety and/or depression symptoms in the past 4 weeks. This is an open-ended question and does not have a scale.
Impact of supervisor's leadership and organizational inclusion on receiving an accommodation and disclosing in the workplace. | 8 weeks
  Supervisors Leader and Organizational Inclusion scales will be used to measure the impact of both on receiving an accommodation or disclosing in the workplace.
  Supervisor Leadership - Min score = 7; Max score = 35 - Higher scores represents more supportive leadership style Organization Inclusion: Min score = 1; Max score = 34 - Higher scores represents a more inclusive and support organization.

SECONDARY OUTCOMES:
Impact of psychoeducation course on comfort level of disclosing a mental health condition in the workplace | 8 weeks
  Participants will be asked about their comfort level disclosing a mental health condition in the workplace in the previous 4 weeks. We will be using a likert scale where 1 equals Very Uncomfortable and 4 equal Very Comfortable. A higher value indicates more comfort disclosing.
Impact of psychoeducation course on rates of disclosure in the workplace | 8 weeks
  Participants will be asked if they have disclosed and to whom they disclosed to in the workplace in the previous 4 weeks. Participants will be provided with a list of people (e.g., family, friends, co-workers) and will be asked to click all that apply. No scales will be used.
Identification of the barriers and facilitators to requesting/receiving workplace accommodations for anxiety and/or depression symptoms | 8 weeks
  Participants will be asked to identify the barriers and facilitators for receiving workplace accommodations in the previous 4 weeks. This is an open-ended questions with no scales.
Feedback on the course structure and content | 1 week
  Participants will provide feedback on the course structure and content so revisions can be made to future versions of the course.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No